CLINICAL TRIAL: NCT05846191
Title: Evaluation of Serum Pentraxin 3 and High Sensitive CRP in Female Patients With Gestational Diabetes Mellitus in Second Trimester of Pregnancy.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mai Mohammed Hosny, Resident doctor, Assiut University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: Evaluation of S.pentraxin3&CRP
Record Dates: First submitted 2023-04-26; First posted 2023-05-06 (Actual); Last update posted 2023-05-06 (Actual); Status verified 2023-04

CONDITIONS: Gestational Diabetes Mellitus in Second Trimester of Pregnancy
Keywords: serum pentraxin 3,high sensitive CRP in female patients with gestational diabetes mellitus

STUDY DESIGN:
Intervention Model Description: Evaluation of serum pentraxin 3 and high sensitive CRP in female patients with gestational diabetes mellitus in second trimester of pregnancy.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- serum pentraxin 3 and high sensitive CRP (Other): female with gestational diabetes mellitus in 2nd trimester
  Interventions: Diagnostic Test: serum pentraxin 3 and high sensitive CRP

INTERVENTIONS:
Diagnostic Test: serum pentraxin 3 and high sensitive CRP — serum pentraxin 3 and high sensitive CRP

SUMMARY:
1. To assess the value of serum Pentraxin-3 and high sensitive CRP in females with normal pregnancy and females with gestational diabetes mellitus in second trimester of pregnancy.
2. To study correlations between serum Pentraxin-3 and High sensitive CRP in gestational diabetes.

DETAILED DESCRIPTION:
Gestational diabetes mellitus (GDM) refers to abnormal glucose metabolism that occurs or is discovered during pregnancy, it can cause multiple poor outcomes and increase maternal and child prevalence and mortality.

GDM can increase the risk of type 2 diabetes mellitus (T2DM) and cardiovascular diseases in pregnant women, and the risk of metabolic disorders in their offspring is high, so it's called a disease that affects two generations.(1) The relationship between maternal hyperglycemia and fetal macrosomia together with other complications has been confirmed.(2) Women with GDM have a higher long-term risk of type 2 diabetes mellitus.(3) Pentraxin 3 (PTX3) and high sensitive CRP are both the acute phase proteins belonging to the pentraxin family but with different biological characteristics, CRP belongs to the short PTX, which is an acute phase protein synthesized by the hepatocytes when the body is stimulated by microbial invasion or tissue damage.(4) PTX3 is a long-chain PTX protein. A variety of tissue cells can produce PTX3 under the stimulation of pro-inflammatory factors, including the endothelial cells, fibroblasts, monocytes, adipocytes, etc.(5,6) There is one study(Changes of serum pentraxin-3 and hypersensitive CRP levels during pregnancy and their relationship with gestational diabetes mellitus , 2019) , that has come to PTX3 and hs-CRP may be related to the pathogenesis of GDM, and they are significantly increased in the second trimester, which provides a new idea for early prevention and treatment of GDM .

ELIGIBILITY:
Inclusion Criteria:

1. Pregnant women.
2. Diagnosed GDM. 3Gestational age >20weeks

Exclusion Criteria:

1. Women with pregestational diabetes .
2. Women with chronic diseases.
3. Twin pregnancy.

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Gender Based: Yes
Enrollment: 90 (Estimated)
Dates: Start 2023-12-05 (Estimated); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-03-10 (Estimated)

PRIMARY OUTCOMES:
Mean different in concentration of serum pentraxin-3 and high sensitive CRP levels in study groups. | 2 years
  female patients with gestational diabetes mellitus in second trimester of pregnancy

REFERENCES:
- [Background] Zhao B, Han X, Meng Q, Luo Q. Early second trimester maternal serum markers in the prediction of gestational diabetes mellitus. J Diabetes Investig. 2018 Jul;9(4):967-974. doi: 10.1111/jdi.12798. Epub 2018 Jan 28. PMID 29288571
- [Background] Dongel I, Gokmen AA, Gonen I, Kaya S. Pentraxin-3 and inflammatory biomarkers related to posterolateral thoracotomy in Thoracic Surgery. Pak J Med Sci. 2019 Mar-Apr;35(2):464-469. doi: 10.12669/pjms.35.2.181. PMID 31086534